CLINICAL TRIAL: NCT06975826
Title: A Comparison Between the Percutaneous Internal Ring Suturing (PIRS) Technique and Laparoscopic Intraperitoneal Purse String Suture Sac Closure Technique in Pediatrics
Brief Title: A Comparison Between Two Laparoscopic Techniques in Management of Inguinal Hernias in Pediatrics
Acronym: Pediatrics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nour eldein Ali Thabet, Assistant lecturer, Advanced Bionics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Laparscopic herniotomy in ped.
Record Dates: First submitted 2025-01-26; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Inguinal Hernia; Pediatrics
Keywords: Laparscopic inguinal herniotomy
MeSH Terms: conditions — Hernia, Inguinal | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laparscopic percutaneous internal ring suturing (PIRS) technique in Management of inguinal hernia (Active Comparator): Use of laparoscopy in Management of inguinal hernia in pediatrics without entering peritoneal cavity
  Interventions: Procedure: Laparscopic percutaneous internal ring suturing (PIRS) technique in Management of inguinal hernia
- Laparoscopic intraperitoneal purse string suture sac closure technique in pediatrics. (Active Comparator): Use of laparoscopy in Management of inguinal hernia in pediatrics through entering peritoneal cavity
  Interventions: Procedure: Laparscopic inguinal herniotomy in pediatrics

INTERVENTIONS:
Procedure: Laparscopic percutaneous internal ring suturing (PIRS) technique in Management of inguinal hernia — Laparscopic percutaneous internal ring suturing (PIRS) technique
  Arms: Laparscopic percutaneous internal ring suturing (PIRS) technique in Management of inguinal hernia
Procedure: Laparscopic inguinal herniotomy in pediatrics — Laparoscopic intraperitoneal purse string suture sac closure technique in pediatrics.
  Arms: Laparoscopic intraperitoneal purse string suture sac closure technique in pediatrics.

SUMMARY:
To compare between the use of the percutaneous internal ring suturing (PIRS) technique and the Laparoscopic intraperitoneal purse-string suture sac closure technique. in pediatrics & evaluate the safety, efficacy feasibility ,operative time ,postoperative pain ,recurrence rate of both approaches.

DETAILED DESCRIPTION:
Inguinal hernia repairs (IHRs) are one of the most common procedures performed by pediatric surgeons around the world. Although the open method remains the most common for pediatric IHR, laparoscopic IHR has increased dramatically between 2009 and 2018. Over a dozen different laparoscopic techniques have been developed .With the rise in popularity of laparoscopic IHR, many researchers have set out to examine the differences in efficacy of open IHR compared with various laparoscopic IHR techniques. However, there are few studies directly comparing different laparoscopic techniques. By determining outcome discrepancies among popular laparoscopic techniques for pediatric IHR, we can help improve surgical techniques, postoperative outcomes, and patient satisfaction.The proposed advantages of the laparoscopic approach include visualization of a contralateral PPV, identification of less common (direct, femoral, pantaloon) hernias ,diminished postoperative pain, more rapid return to normal function, and improved cosmesis. Two laparoscopic techniques that have gained popularity among pediatric surgeons in the past decade, the percutaneous internal ring suturing (PIRS) technique and Laparoscopic intraperitoneal purse string suture sac closure technique.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 1month to 18 years. 2. Denovo Inguinal Hernias. 3. Uncomplicated Inguinal Hernias.

Exclusion Criteria:

* 1. Complicated Inguinal Hernia 2. Age more than 18 Years 3. cases inwhich laparoscopic surgery is contraindicated 4. cases with collagen disease. 5. Recurrent Inguinal Hernia.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-26 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Operative time in both approaches | baseline
  time from start of operation to the end

CONTACTS AND LOCATIONS:
Overall Officials: Almoataz Ahmed Eltayeb, Study Director